CLINICAL TRIAL: NCT00264121
Title: The Incidence of Congenital Undescended Testis Among Dutch Infants in the Medical Centre Alkmaar
Brief Title: The Incidence of Congenital Undescended Testis Among Dutch Infants
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical Center Alkmaar (Other)
Other Study IDs: P05.0318L
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Undescended Testis
Keywords: congenital, high scrotal
MeSH Terms: conditions — Cryptorchidism

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to determine the incidence of congenital undescended testis of mature boys, at one year of age, born in the Medical Centre Alkmaar (MCA).

DETAILED DESCRIPTION:
The position of the testes of mature boys will be registered at birth and boys with a high-scrotal, non-scrotal or dubious position of the testis/ testes will be followed up (till the age of one year).

ELIGIBILITY:
Inclusion Criteria:

* mature newborns (>/= 37 weeks)
* born in the Medical Centre Alkmaar

Exclusion Criteria:

* premature newborns (< 37 weeks)

Max Age: 1 Year | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3000 (Estimated)
Dates: Start 2005-06; Study Completion 2008-06

CONTACTS AND LOCATIONS:
Overall Officials: W WM Hack, PhD, Study Director — Department of Pediatrics, Medical Centre Alkmaar
Locations (1):
- Medical Center Alkmaar (MCA), Alkmaar, North Holland, Netherlands